CLINICAL TRIAL: NCT02232581
Title: Randomised, Double Blind, Placebo-controlled Dose Ranging Trial to Determine the Antiviral Activity and Safety of Alovudine in Nucleoside-experienced HIV-infected Subjects Experiencing Virologic Failure
Brief Title: Study to Determine the Antiviral Activity and Safety of Alovudine in Nucleoside-experienced HIV-infected Subjects Experiencing Virologic Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1211.1
Record Dates: First submitted 2014-09-04; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

ARMS (4):
- Alovudine - low (Experimental)
  Interventions: Drug: Alovudine - low; Drug: Placebo
- Alovudine - medium (Experimental)
  Interventions: Drug: Alovudine - medium; Drug: Placebo
- Alovudine - high (Experimental)
  Interventions: Drug: Alovudine - high
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alovudine - low
  Arms: Alovudine - low
Drug: Alovudine - medium
  Arms: Alovudine - medium
Drug: Alovudine - high
  Arms: Alovudine - high
Drug: Placebo
  Arms: Alovudine - low; Alovudine - medium; Placebo

SUMMARY:
The primary objective was to determine the mean change in HIV viral load from baseline to Week 4 compared with placebo after 4 weeks of treatment in highly experienced HIV-infected patients.

Secondary objectives were to determine (1) the tolerability, hematologic and hepatic safety of different doses of alovudine and (2) the effect of baseline nucleoside genotypic susceptibility on virologic response after 4 weeks of alovudine administration

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any trial procedure
* HIV-1 infected males or females ≥18 years of age
* Screening genotypic resistance report indicating two or more of the following nucleoside reverse transcriptase inhibitors (NRTI) resistance mutations: 41, 67, 70, 210 and 215
* Stable NRTI regimen without stavudine and zidovudine for at least 6 weeks before screening and stable antiretroviral (ARV) background treatment for 3 months before screening
* HIV-1 viral load ≥1000 copies/mL and <75,000 copies/mL at screening
* Change in viral load between previous test within 3 months before screening, using local laboratory for routine tests, and screening test was <1.0 log10 copies/mL
* Acceptable medical history, as assessed by the investigator
* Current stable ARV medication regimen between screening (Visit 1) and Visit 2

Exclusion Criteria:

* ARV medication naïve
* Patients on recent drug holiday, defined as off ARV medications for at least 7 consecutive days within the previous 3 months
* Female patients of child-bearing potential who :

  * have a positive serum pregnancy test
  * are breast feeding,
  * are planning to become pregnant, or
  * are not willing to use a barrier method of contraception
* Prior alovudine use
* Use of investigational medications within 30 days before study entry or during the trial
* Use of immunomodulatory drugs within 3 months before study entry or during the trial (e.g. interferon, cyclosporine, hydroxyurea, interleukin-2)
* Current use of rifampin, rifabutine, isoniazid, pyrazinamide, stavudine, zidovudine, ganciclovir, chronic use of hepatotoxic drugs, anti-tumour therapy or probenecid
* Laboratory values:

  * Neutrophils of Grade 2 or greater abnormality
  * Hemoglobin of Grade 2 or greater abnormality
  * Platelets: Grade 2 or greater abnormality
  * Creatinine of ≥1.25 Upper limit of the normal (ULN)
  * Lipase of Grade 1 or greater abnormality
  * Alanine aminotransaminase (ALT) or Aspartate aminotransaminase (AST) of Grade 2 or greater abnormality
  * Direct bilirubin of Grade 1 or greater abnormality
* CD4 ≤50 cells/mm3
* Hepatitis B (+HBsAg or +HBcAB) or C +Hepatitis C virus (+HCV AB ) co-infection, chronic hepatitis, on-going hepatitis or pancreatitis
* Any new or active AIDS-defining event within 30 days before study entry
* Inability to adhere to the requirements of the protocol, including active substance abuse as assessed by the investigator
* In the opinion of the investigator, likely survival of less than 6 months because of underlying disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-04; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Mean change in HIV viral load measured from plasma samples | Up to 4 weeks after drug administration

SECONDARY OUTCOMES:
Percentage of virologic responders per treatment arm | Up to 4 weeks after drug administration
Proportion of patients experiencing a change of viral load | Up to 4 weeks after drug administration
  viral load of ≥1 log10 from baseline to Week 4
Mean change in CD4+ cell count | Up to 4 weeks after drug administration
Percentage of 0.5 virologic responders per treatment arm | Up to 4 weeks after drug administration
Percentage of load responders per treatment arm | Up to 4 weeks after drug administration
Percentage of 0.7 to 0.9 virologic responders per treatment arm | Up to 4 weeks after drug administration
Number of patients with adverse events | Up to 4 weeks after drug administration
Number of patients with laboratory test abnormalities and with respect to Division of AIDS (DAIDS) grading | Up to 4 weeks after drug administration
Number of patients with serious adverse events | Up to 4 weeks after drug administration
Number of patients who discontinued due to adverse event | Up to 4 weeks after drug administration
Mean change in CD8+ cell count | Up to 4 weeks after drug administration
Number of patients with abnormal changes in laboratory parameters | Up to 4 weeks after drug administration